CLINICAL TRIAL: NCT00061802
Title: A Randomized, Double Blind Study to Evaluate the Efficacy and Safety of Two Atypical Antipsychotics vs. Placebo in Patients With an Acute Exacerbation of Either Schizophrenia or Schizoaffective Disorder
Brief Title: Efficacy and Safety of Two Atypical Antipsychotics vs. Placebo in Patients With an Acute Exacerbation of Either Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002890
Record Dates: First submitted 2003-06-04; First posted 2003-06-05 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Quetiapine Fumarate

INTERVENTIONS:
Drug: risperidone, quetiapine

SUMMARY:
A study to evaluate the efficacy and safety of two atypical antipsychotics vs. placebo in patients with an acute exacerbation of either schizophrenia or schizoaffective disorder

DETAILED DESCRIPTION:
This study was intended to compare the efficacy and safety of risperidone, quetiapine, and placebo in the treatment of patients with acute exacerbations of schizophrenia or schizoaffective disorder. The primary tested hypothesis was a comparison of the efficacy of risperidone and quetiapine (active combined group) to placebo. Other a priori hypotheses tested included comparison of the onset of antipsychotic effect of risperidone to quetiapine and placebo, and to evaluate the efficacy, safety, and cost of risperidone compared with quetiapine in the treatment of subjects with an acute exacerbation of schizophrenia or schizoaffective disorder.

During the first phase of the study (15 days), patients randomized to risperidone were titrated from 1 mg to 4 mg or from 1 mg to 6 mg per day, depending on body weight. Patients randomized to quetiapine were titrated from 50 mg to 400 mg or from 50 mg to 600 mg per day, depending on body weight. Based on investigators determination of patient clinical response, patients in the quetiapine group could be titrated to a maximum of 600 mg or 800 mg per day depending on body weight.

During the second phase of the study (days 15 - 42), patients continue to take the dose of study medication taken in the first phase, but additional psychotropic medication could be added as clinically necessary to control symptoms in patients who remained sufficiently symptomatic (defined as a certain minimum value on a clinical global severity scale.)

ELIGIBILITY:
Current diagnosis of an acute exacerbation of either schizophrenia or schizoaffective disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2003-06; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of combined risperidone and quetiapine groups versus placebo based on change in psychotic symptoms scale from baseline to two weeks.

SECONDARY OUTCOMES:
Comparison of response rates based on proportion of patients in each study group that reach a predetermined percent decrease in psychotic symptom score at two weeks.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - San Diego, California
  - Hoffman Est, Illinois
  - Lake Charles, Louisiana
  - Jackson, Mississippi
  - Visakhapatnam, Missouri
  - The Bronx, New York
  - Oklahoma City, Oklahoma
- India (4):
  - Aurangabad
  - New Delhi
  - Orange
  - San Diego
- Romania (2):
  - Lucknow
  - Richmond

REFERENCES:
- [Result] Gharabawi GM, Greenspan A, Rupnow MF, Kosik-Gonzalez C, Bossie CA, Zhu Y, Kalali AH, Awad AG. Reduction in psychotic symptoms as a predictor of patient satisfaction with antipsychotic medication in schizophrenia: data from a randomized double-blind trial. BMC Psychiatry. 2006 Oct 20;6:45. doi: 10.1186/1471-244X-6-45. PMID 17054789